CLINICAL TRIAL: NCT06302179
Title: Risk Factors of Venous Thromboembolism After Colorectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 140-14/24
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Venous Thromboembolism
Keywords: colorectal cancer surgery; thromboprophylaxis
MeSH Terms: conditions — Colorectal Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of our study is to find frequency and identify risk factors for venous thromboembolism development in patients who underwent surgery for colorectal cancer. There were 137 patients enrolled in our retrospective observational cohort study. Included patients were operated for incisional hernia in Saveljev University Surgery Clinic from January 2016 to December 2017. Compression duplex ultrasound of lower legs veins was performed in 2-14 days after surgery for all participants. The primary endpoint was the occurrence of the venous thromboembolism event, including pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

operated for incisional hernia in Saveljev University Surgery Clinic. No Exclusion Criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Venous Thromboembolism | was performed with median 4 days (min 2 day, max 14 days, interquartile range 2-5 days) after surgery
  Screening ultrasound in the postoperative period was aimed at looking for signs of deep vein thrombosis. The imaged vessels included the common femoral, great saphenous, superficial femoral, deep femoral, popliteal, posterior tibial, and peroneal veins of both lower extremities. The presence of a thrombotic process in the vein was evidenced by the rigidity of its walls during compression by the sensor, the presence of hyperechoic inclusions, and the impossibility of visualizing blood flow during color mapping.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia